CLINICAL TRIAL: NCT05190185
Title: A Clinical Trial of TAA06 Injection in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-TAA06-001
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Malignant Melanoma, Lung Cancer, or Colorectal Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAA06 injection (Experimental): T cell injection targeting B7-H3 chimeric antigen receptor
  Interventions: Biological: TAA06 injection

INTERVENTIONS:
Biological: TAA06 injection — The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be treated with 1×106~1×108 CAR-T/kg. And the subjects will be administered once.

SUMMARY:
B7-H3 (also known as CD276) is widely expressed on the surface of a variety of malignancies solid tumors, while it rarely or even doesn't express on normal tissues. Therefore, B7-H3 is an ideal target for chimeric antigen receptor (CAR) T cells therapy. TAA06 injection is a CAR T injection targeting B7-H3. This is a phase I clinical study with the primary objective of evaluating the safety and tolerability of TAA06 injection in subjects with TAA06-positive advanced solid tumors. The secondary objectives are as follows: to evaluate the distribution, proliferation and persistence of B7-H3-targeted CAR T cells after injection of TAA06 in subjects; to preliminarily evaluate the efficacy of TAA06 injection in subjects with TAA06-positive advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 18 to 70 years old (inclusive), male or female;
* (2) Expected survival time ≥ 12 weeks;
* (3) ECOG performance status of 0-1;
* (4) It is clearly diagnosed by pathology to be any of the following tumor types: malignant melanoma, lung cancer or colorectal cancer, and the positive rate of TAA06 expression in tumor tissues is ≥1% after immunohistochemical detection;
* (5) Subjects whose standard treatment methods are ineffective (eg: relapse after surgery, disease progress after treatment with chemotherapy, radiotherapy or targeted drugs);
* (6) According to the curative effect evaluation standard for solid tumors (RECIST 1.1), at least one measurable lesion (the longest diameter of the solid lesion ≥ 10mm, or the short diameter of the lymph node lesion ≥ 15mm);
* (7) The main organ function is normal (white blood cell count ≥3×109/L, neutrophil count ≥1.5×109/L, hemoglobin ≥8.5g/dL, platelet count ≥80×109/L, lymphocyte count at 1×109/L (inclusive) ~ 4×109/L (inclusive));
* (8) Liver and kidney function, heart and lung function meet the following criteria:

  1. Urea (Urea) and serum creatinine≤1.5×ULN;
  2. Left ventricular ejection fraction ≥50%;
  3. Baseline blood oxygen saturation ≥ 94%;
  4. Total bilirubin≤1.5×ULN; ALT and AST≤2.5×ULN;
* (9) The subjects or his legal representative can fully understand the significance and risks of this trial and has signed informed consents.

Exclusion Criteria:

* (1) Subjects with a history of immunodeficiency or autoimmune diseases (including but not limited to rheumatoid joint disease, systemic lupus erythematosus, vasculitis, multiple sclerosis, insulin-dependent diabetes, etc.); with graft-versus-host disease (GVHD) , Or those who need to use immunosuppressive agents;
* (2) Subjects with other type of malignant tumors within 5 years prior to screening;
* (3) Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA titer detection not within the normal reference range; positive for hepatitis C virus (HCV) antibody and peripheral blood hepatitis C virus (HCV) RNA; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis test;
* (4) Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmia;
* (5) Unstable systemic diseases judged by the investigator: including but not limited to serious liver, kidney or metabolic diseases requiring drug treatment;
* (6) Within 7 days prior to screening, there are active or uncontrollable infections requiring systemic therapy (except for mild genitourinary infection and upper respiratory tract infection);
* (7) Pregnant or lactating women, and female subjects who plan to become pregnant within 1 year after cell infusion or male subjects whose partners plan to become pregnant within 1 year after cell infusion;
* (8) Subjects who have received CAR-T therapy or other gene-modified cell therapy prior to screening;
* (9) Subjects who are receiving systemic steroid therapy within 7 days prior to screening or need long-term use of systemic steroid therapy during treatment as judged by the investigator (except for inhalation or topical use);
* (10) Subjects with more than a moderate amount of ascites, or after conservative medical treatment (such as diuresis, sodium restriction, excluding ascites drainage) for 2 weeks, the ascites still shows a progressive increase;
* (11) Conditions not eligible for cell preparation as judged by the investigator;
* (12) Other conditions considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety after B7-H3 chimeric antigen receptor T cells infusion (Safety) | 3 months
  Incidence and treatment-relativity of adverse events assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
To evaluate anti-tumor activity (overall response rate) | 6 months
  Rate of participants achieving a complete response (CR) or partial response (PR).
To evaluate anti-tumor activity (disease control rate) | 3 months
  Rate of participants achieving a complete response (CR) or partial response (PR) or stable disease (PD).
To evaluate anti-tumor activity (duration of response) | About 2 years
  Defined as the time from the first tumor assessment of CR or PR to the first assessment of disease progression (PD) or death from any cause.
To evaluate anti-tumor activity (Progression Free Survival) | About 2 years
  Defined as the time from the date of study enrollment to the time when the investigator judges that imaging disease progression or death from any cause occurs.
To evaluate anti-tumor activity (overall survival) | About 2 years
  Defined as the time from start of the random beginning to death (due to any cause).

CONTACTS AND LOCATIONS:
Locations (1):
- PersonGen BioTherapeutics(Suzhou) Co., Ltd., Suzhou, Jiangsu, China